CLINICAL TRIAL: NCT00753844
Title: Tumor Vaccine Therapy Against Advanced Esophageal Cancer Using HLA-A*2402 Restricted Epitope Peptides Drived From URLC10
Brief Title: Human Leukocyte Antigen (HLA) - A*2402 Restricted Peptide Vaccine Therapy in Patients With Advanced Esophageal Cancer
Status: Completed | Phase: Phase 1 | Type: Interventional
Sponsor: Kinki University (Other)
Collaborators: Human Genome Center, Institute of Medical Science, University of Tokyo (Other)
Responsible Party: Principal Investigator, Hajime Ishikawa, department of surgery, Kinki University
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: 18-29
Record Dates: First submitted 2008-09-16; First posted 2008-09-17 (Estimated); Last update posted 2012-04-06 (Estimated); Status verified 2012-04

CONDITIONS: Esophageal Cancer
Keywords: peptide vaccine; URLC10
MeSH Terms: conditions — Esophageal Neoplasms | interventions — LY6K protein, human

INTERVENTIONS:
Biological: URLC10 — Biological: URC10 Patients will be vaccinated once in one week to the eighth vaccine and will be vaccinated once in two weeks from the ninth vaccine. On each vaccination day, the URLC10 peptide (1mg) mixed with Montanide ISA 51 will be administered by endodermic injection.

SUMMARY:
The purpose of this study it to evaluate the safety and immune response of peptides (URLC10) emulsified with Montanide ISA51 in treating patients with unresectable, advanced or recurrent esophageal cancer.

DETAILED DESCRIPTION:
URLC10 have been identified as cancer specific molecules especially in non small cell lung cancer using genome-wide expression profile analysis by cDNA microarray technique. In a prior study, it has been shown that URLC10 are upregulated in human esophageal tumors. The investigators identified that peptides derived from these proteins significantly induce the effective tumor specific CTL response in vitro. According to these findings, in this trial, we evaluate the safety, immunological and clinical response of URLC10 peptide. Patients will be vaccinated once in one week to the eighth vaccine and will be vaccinated once in two weeks from the ninth vaccine. On each vaccination day, the URLC10 peptide (1mg) mixed with Montanide ISA 51 will be administered by endodermic injection

ELIGIBILITY:
Inclusion Criteria:

1. Patients must have Advanced or recurrent esophageal cancer, and treatment has failed, or in the situation where effective therapy is not available, or has been refused due to severe adverse effects of chemotherapy
2. WHO performance status of 0 to 2
3. Age ≥ 20 years, ≤80 years
4. The patient does not need to have a measurable disease, but must have a disease that an effect judgment is possible
5. Passing from previous treatment more than two weeks. Passing from radiation therapy more than four weeks.
6. Expected survival of at least 3 months
7. WBC≥ 1,500/mm³ WBC≤ 15,000/mm³ Platelet count ≥ 50,000/mm³ Total bilirubin ≤ 3 x the institutional normal upper limits AST, ALT ≤ 3 x the institutional normal upper limits Creatinine ≤ 3 x the institutional normal upper limits
8. Patients must be HLA-A2402
9. Able and willing to give valid written informed consent

Exclusion Criteria:

1. Pregnancy, Promise of the pregnancy, Hope of the pregnancy, Breastfeeding
2. Serious infections requiring antibiotics
3. Concurrent treatment with steroids or immunosuppressing agent
4. Disease to the central nervous system
5. Decision of unsuitableness by principal investigator or physician-in-charge

Ages: 20 Years to 80 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 7 (Actual)
Dates: Start 2006-11; Primary Completion 2009-06 (Actual); Study Completion 2009-07 (Actual)

PRIMARY OUTCOMES:
Safety(Phase I:toxicities as assessed by NCI CTCAE version3) | 28 days after beginning protocol

SECONDARY OUTCOMES:
efficacy(Feasibility as evaluated by RECIST) | 28 days after beginning protocol
evaluate immunological responses | 28 days after beginning protocol

CONTACTS AND LOCATIONS:
Locations (1):
- department of surgery, Kinki University, Sayama, Osaka, Japan